CLINICAL TRIAL: NCT02068352
Title: A Phase 2 Multi-center, Randomized, Double-blind, Vehicle-controlled, Three-arm, Parallel Group Study to Assess the Safety, Tolerability, and Efficacy of Topical OPA-15406 Ointment, in Subjects With Mild/Moderate Atopic Dermatitis
Brief Title: A Study to Evaluate the Effectiveness and Safety of Topical OPA-15406 Ointment to Treat Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 271-12-205; 2013-003899-12 (EudraCT Number)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis, Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — difamilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.3% OPA-15406 (Experimental): OPA-15406 0.3% ointment was applied topically twice daily (BID) to the selected treatment area(s) at approximately 12-hour intervals for 8 weeks.
  Interventions: Drug: OPA-15406
- 1% OPA-15406 (Experimental): OPA-15406 1% ointment was applied topically BID to the selected treatment area(s) at approximately 12-hour intervals for 8 weeks.
  Interventions: Drug: OPA-15406
- Vehicle Ointment (Placebo Comparator): OPA-15406 1%-matching placebo (vehicle ointment) was applied topically BID to the selected treatment area(s) at approximately 12-hour intervals for 8 weeks.
  Interventions: Drug: Vehicle ointment

INTERVENTIONS:
Drug: OPA-15406 — OPA-15406 topical ointment
  Arms: 0.3% OPA-15406; 1% OPA-15406
Drug: Vehicle ointment — OPA-15406 1%-matching placebo topical ointment
  Arms: Vehicle Ointment

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of 2 concentrations of OPA-15406 compared to vehicle in participants with atopic dermatitis (AD).

DETAILED DESCRIPTION:
AD is a disease mainly characterized by pruritic eczema, and those with the disease experience repeated exacerbations and remissions. Therapeutic guidelines for the disease, currently being developed in many countries, all recognize AD as chronic eczema that is accompanied by the physiological dysfunction of the skin and in which inflammation is caused by various nonspecific stimuli or specific allergens. OPA 15406 is a type-4 phosphodiesterase (PDE4) inhibitor. PDE4 inhibitors are thought to be useful for allergic inflammatory diseases. This is a Phase 2 dose ranging study to evaluate the efficacy of two concentrations of OPA 15406 ointment compared to vehicle, when administered topically twice daily in participants with mild to moderate AD.

ELIGIBILITY:
Inclusion Criteria:

* Participants 10-70 years of age
* Diagnosis of AD
* History of AD for at least 3 years
* AD affecting greater than or equal to 5% and less than or equal to 40% of total body surface area (BSA) at Baseline
* Investigator's Global Assessment of Disease Severity score of 2 (mild) or 3 (moderate) in the selected treatment area(s)

Exclusion Criteria:

* Contact or atopic dermatitis flare within 28 days of the Baseline (Day 1) visit.
* Concurrent diseases/conditions and history of other diseases/conditions in the selected treatment area(s) that may have an impact on the study assessments.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-06-20 (Actual); Primary Completion 2015-01-28 (Actual); Study Completion 2015-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (20):
  - Los Angeles, California
  - San Diego, California
  - Denver, Colorado
  - Orange Park, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Arlington Heights, Illinois
  - Carmel, Indiana
  - Ann Arbor, Michigan
  - Verona, New Jersey
  - Albuquerque, New Mexico
  - Stony Brook, New York
  - High Point, North Carolina
  - Portland, Oregon
  - Austin, Texas
  - College Station, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Spokane, Washington
- Australia (5):
  - Phillip, Australian Capital Territory
  - Kogarah, New South Wales
  - Woolloongabba, Queensland
  - Hectorville, South Australia
  - Fremantle, Western Australia
- Poland (5):
  - Katowice
  - Krakow
  - Lodz
  - Warsaw
  - Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 30 investigative sites in Australia, Poland, and the United States from 20 June 2014 to 28 January 2015.
Pre-assignment Details: Participants with mild/moderate atopic dermatitis were randomized in 1:1:1 ratio to receive OPA 15406 (3% w/w, 1% w/w) and matching placebo. Participants had screening evaluations between 30 and 2 days before entering the 8-week treatment phase.
Period: Overall Study
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
Started | 41 | 43 | 37
Completed | 31 | 35 | 28
Not Completed | 10 | 8 | 9
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Adverse Event | 4 | 2 | 7
Not completed — Participant met (Protocol Specified) Withdrawal Criteria | 0 | 1 | 0
Not completed — Participant Withdrew Consent to Participate | 6 | 3 | 1
Not completed — Protocol Deviation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Efficacy Sample included all participants who were randomized and received at least one dose of investigational medicinal product (IMP).
Groups:
- 0.3% OPA-15406: OPA-15406 0.3% ointment was applied topically BID to the selected treatment area(s) at approximately 12-hour intervals for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment | Total
Number analyzed (Participants) | 41 | 43 | 37 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (15.2) | 34.1 (16.5) | 32.2 (15.6) | 34.3 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 23 | 72
  Male | 14 | 21 | 14 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 7 | 18
  Not Hispanic or Latino | 37 | 36 | 30 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 3
  Black or African American | 14 | 11 | 5 | 30
  White | 24 | 30 | 28 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Success in the Overall Investigator's Global Assessment of Disease Severity (IGA) Score at Week 4 [Using Non-responder Imputation or Last Observation Carried Forward (LOCF)]
Description: The IGA evaluation was performed by a certified rater. The IGA score, used to assess the overall disease severity, consists of a 6-point severity scale from clear to very severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease, and 5 = very severe disease). The IGA uses clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines for the overall severity assessment. The IGA assessment was performed for the overall selected treatment area(s): overall percentage body surface area to be treated and additionally for the target lesion. Success was defined as a score of 0 or 1 with at least a 2-grade reduction from Baseline. Participants without IGA score at Week 4 were treated as non-responders. In the sensitivity analysis, missing IGA score at Week 4 was imputed using LOCF method first and the success was defined based on the imputed IGA score.
Time Frame: Week 4
Population: Efficacy Sample included all participants who were randomized and received at least one dose of IMP. Number analyzed is the number of participants meeting responder criteria defined as an IGA score of 0 or 1 and at least 2-grade reduction from Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
Number analyzed (Participants) | 41 | 43 | 37
percentage of participants
  Non-responders | 14.63 | 20.93 | 2.70
  LOCF: number analyzed (Participants) | 40 | 43 | 37
  LOCF | 15.00 | 20.93 | 2.70
Statistical Analysis 1: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0690, Cochran-Mantel-Haenszel — P-value was derived using Cochran-Mantel-Haenszel (CMH) test stratified by age group (< 18 or ≥ 18) and region; Mean Difference = 11.93, 95% CI 2-sided [-0.08 to 23.95]
Statistical Analysis 2: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0165, Cochran-Mantel-Haenszel — P-value was derived using CMH test stratified by age group (< 18 or ≥ 18) and region; Mean Difference = 18.23, 95% CI 2-sided [4.99 to 31.46]
Statistical Analysis 3: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0617, Cochran-Mantel-Haenszel — P-value was derived using CMH test stratified by age group (< 18 or ≥ 18) and region; Mean Difference = 12.30, 95% CI 2-sided [0.06 to 24.53]

2. Secondary Outcome: Change From Baseline in Overall IGA Score at Week 4 [Using Mixed Model Repeated Measures (MMRM) Analysis]
Description: The IGA evaluation was performed by a certified rater. The IGA allows for an assessment of overall disease severity at a given time point, and it consists of a 6-point severity scale from clear to very severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease, and 5 = very severe disease). The IGA uses clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines for the overall severity assessment. The IGA assessment was performed for the overall selected treatment area(s): overall percentage body surface area to be treated and additionally for the target lesion. A negative change from Baseline indicates improvement in overall IGA score.
Time Frame: Baseline, Week 4
Population: Efficacy Sample included all randomized participants who received at least one dose of study treatment. Overall number analyzed is the number of participants with non-missing assessment at a specific visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
Number analyzed (Participants) | 35 | 40 | 29
score on a scale | -0.56 (0.14) | -0.55 (0.13) | -0.09 (0.15)
Statistical Analysis 1: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0128, Mixed Models Analysis; MMRM with fixed effects of treatment, region, visit, age group, and interaction of treatment by visit as terms, Baseline score as a covariate; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.84 to -0.10]
Statistical Analysis 2: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0134, Mixed Models Analysis; MMRM with fixed effects of treatment, region, visit, age group, interaction of treatment by visit, Baseline score as a covariate; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.81 to -0.10]

3. Secondary Outcome: Change From Baseline in Overall IGA Score at Week 4 [Using Last Observation Carried Forward (LOCF) Analysis]
Description: The IGA allows for an assessment of overall disease severity at a given time point, and it consists of a 6-point severity scale from clear to very severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease, and 5 = very severe disease). The IGA uses clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines for the overall severity assessment. Missing overall IGA scores at Week 4 were imputed using LOCF method. A negative change from Baseline indicates improvement in overall IGA score.
Time Frame: Baseline, Week 4
Population: Efficacy Sample included all participants who were randomized and received at least one dose of IMP. Overall number analyzed is the number of participants with non-missing assessment at a specific visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
Number analyzed (Participants) | 40 | 43 | 37
score on a scale | -0.54 (0.15) | -0.54 (0.14) | -0.04 (0.15)
Statistical Analysis 1: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0048, ANCOVA; Analysis of covariance (ANCOVA) model with treatment, region, age group as terms, and Baseline score as a covariate for change from Baseline; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.85 to -0.16]
Statistical Analysis 2: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0045, ANCOVA; ANCOVA model with treatment, region, age group as terms, and Baseline score as a covariate for change from Baseline; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.84 to -0.16]

4. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An serious adverse event (SAE) was defined as any event which resulted in death, was life-threatening, was a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, required in-patient hospitalization or prolonged hospitalization, was a congenital anomaly/birth defect, or was another medically significant event.
Time Frame: From signing of informed consent through Week 8
Population: Safety Sample included all participants who received at least one dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
Number analyzed (Participants) | 41 | 43 | 37
percentage of participants
  Participants With Treatment Site AEs | 26.8 | 11.6 | 18.9
  Participants With Treatment-emergent AEs (TEAEs) | 58.5 | 41.9 | 54.1
  Participants With Serious TEAEs | 4.9 | 4.7 | 0.0
  Participants With Severe TEAEs | 12.2 | 4.7 | 8.1
  Participants With Severe Treatment Site TEAEs | 4.9 | 0.0 | 5.4

5. Other Pre Specified Outcome: Percentage of Participants With Success in the Overall IGA Score at Week 8 (Using Non-responder Imputation or LOCF Imputation)
Description: IGA evaluation was performed by a certified rater. The IGA consists of a 6-point severity scale from clear to very severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease, and 5 = very severe disease). The IGA uses clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines for the overall severity assessment. The IGA assessment was performed for the overall selected treatment area(s): overall percentage body surface area to be treated and additionally for the target lesion. Success was defined as a score of 0 or 1 with at least a 2-grade reduction from Baseline. In the primary analysis, participants without IGA score available at Week 8 were treated as non-responders. In the sensitivity analysis, the missing IGA score at Week 8 was imputed using LOCF method first and the success was defined based on the imputed IGA score.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
Number analyzed (Participants) | 41 | 43 | 37
percentage of participants
  Non-responders | 17.07 | 16.28 | 10.81
  LOCF: number analyzed (Participants) | 40 | 43 | 37
  LOCF | 20.00 | 20.93 | 10.81
Statistical Analysis 1: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.4173, Cochran-Mantel-Haenszel — P-value was derived using CMH test stratified by age group (< 18 or ≥ 18) and region; Mean Difference (Final Values) = 6.26, 95% CI 2-sided [-8.99 to 21.52]
Statistical Analysis 2: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.4895, Cochran-Mantel-Haenszel — P-value was derived using CMH test stratified by age group (< 18 or ≥ 18) and region; Mean Difference (Final Values) = 5.47, 95% CI 2-sided [-9.43 to 20.36]
Statistical Analysis 3: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.2677, Cochran-Mantel-Haenszel — P-value was derived using CMH test stratified by age group (< 18 or ≥ 18) and region; Mean Difference (Final Values) = 9.19, 95% CI 2-sided [-6.74 to 25.12]
Statistical Analysis 4: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.2319, Cochran-Mantel-Haenszel — P-value was derived using CMH test stratified by age group (< 18 or ≥ 18) and region; Mean Difference (Final Values) = 10.12, 95% CI 2-sided [-5.63 to 25.87]

6. Other Pre Specified Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) Score (Using MMRM Analysis)
Description: The EASI evaluation assesses the extent of disease at 4 body sites and measures 4 clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each on a scale from 0 (no disease) to 3 (very severe). The EASI scale allows for a maximum score of 72. The EASI assessment was performed on overall body. A negative change from Baseline indicates improvement in EASI score.
Time Frame: Baseline, Weeks 4 and 8
Population: Efficacy Sample included all participants who were randomized and received at least one dose of IMP. Number analyzed is the number of participants with non-missing assessment at a specific visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
Number analyzed (Participants) | 41 | 43 | 37
score on a scale
  Change at Week 4: number analyzed (Participants) | 35 | 40 | 29
  Change at Week 4 | -2.21 (0.85) | -3.19 (0.80) | -1.10 (0.90)
  Change at Week 8: number analyzed (Participants) | 31 | 35 | 28
  Change at Week 8 | -2.60 (0.90) | -3.47 (0.86) | -1.57 (0.95)
Statistical Analysis 1: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.3213, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Mean Difference (Final Values) = -1.11, 95% CI 2-sided [-3.33 to 1.11]
Statistical Analysis 2: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0594, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Mean Difference (Final Values) = -2.09, 95% CI 2-sided [-4.27 to 0.08]
Statistical Analysis 3: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.396, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-3.43 to 1.37]
Statistical Analysis 4: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.1135, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Mean Difference (Final Values) = -1.90, 95% CI 2-sided [-4.26 to 0.46]

7. Other Pre Specified Outcome: Change From Baseline in EASI Score (Using LOCF Analysis)
Description: as for outcome 6
Time Frame: Baseline, Weeks 4 and 8
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
Number analyzed (Participants) | 41 | 43 | 37
score on a scale
  Change at Week 4: number analyzed (Participants) | 40 | 43 | 37
  Change at Week 4 | -2.00 (0.91) | -3.07 (0.87) | -0.51 (0.92)
  Change at Week 8: number analyzed (Participants) | 40 | 43 | 37
  Change at Week 8 | -2.42 (1.01) | -3.36 (0.96) | -1.00 (1.02)
Statistical Analysis 1: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.1703, ANCOVA; ANCOVA model with treatment, region, age group as terms, and Baseline score as a covariate for change from Baseline; Mean Difference (Final Values) = -1.49, 95% CI 2-sided [-3.63 to 0.65]
Statistical Analysis 2: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0176, ANCOVA; ANCOVA model with treatment, region, age group as terms, and Baseline score as a covariate for change from Baseline; Mean Difference (Final Values) = -2.56, 95% CI 2-sided [-4.67 to -0.45]
Statistical Analysis 3: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.2381, ANCOVA; ANCOVA model with treatment, region, age group as terms, and Baseline score as a covariate for change from Baseline; Mean Difference (Final Values) = -1.41, 95% CI 2-sided [-3.78 to 0.95]
Statistical Analysis 4: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.047, ANCOVA; ANCOVA model with treatment, region, age group as terms, and Baseline score as a covariate for change from Baseline; Mean Difference (Final Values) = -2.36, 95% CI 2-sided [-4.68 to -0.03]

8. Other Pre Specified Outcome: Change From Baseline in Visual Analog Scale (VAS) Score for Pruritus (Using MMRM Analysis)
Description: At each evaluation, the participants were asked to record their current pruritus intensity over their body overall, not just within the selected treatment areas[s] (i.e., intensity over the last 24 hours) on a horizontal 100-mm line marked as "No itch" on the left end and "Worst imaginable itch" on the right end. The VAS assessment was performed on the overall impression of itch on the body and not just for the selected treatment area(s) or for the target lesion. A negative change from Baseline indicates improvement in VAS score.
Time Frame: Baseline, Weeks 4 and 8
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
Number analyzed (Participants) | 41 | 43 | 37
units on scale
  Change at Week 4: number analyzed (Participants) | 35 | 40 | 29
  Change at Week 4 | -6.27 (4.67) | -16.71 (4.40) | -4.87 (4.96)
  Change at Week 8: number analyzed (Participants) | 31 | 35 | 28
  Change at Week 8 | -10.98 (5.12) | -20.71 (4.85) | -7.30 (5.44)
Statistical Analysis 1: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.8196, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Mean Difference (Final Values) = -1.40, 95% CI 2-sided [-13.5 to 10.7]
Statistical Analysis 2: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0503, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Mean Difference (Final Values) = -11.83, 95% CI 2-sided [-23.69 to 0.02]
Statistical Analysis 3: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.5902, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Mean Difference (Final Values) = -3.68, 95% CI 2-sided [-17.22 to 9.85]
Statistical Analysis 4: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0482, Mixed Models Analysis; [statistical method as in outcome 2, analysis 2]; Mean Difference (Final Values) = -13.42, 95% CI 2-sided [-26.73 to -0.11]

9. Other Pre Specified Outcome: Change From Baseline in VAS for Pruritus (Using LOCF Analysis)
Description: as for outcome 8
Time Frame: Baseline, Weeks 4 and 8
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
Number analyzed (Participants) | 41 | 43 | 37
units on a scale
  Change at Week 4: number analyzed (Participants) | 40 | 43 | 37
  Change at Week 4 | -4.05 (4.92) | -14.59 (4.64) | -3.05 (4.96)
  Change at Week 8: number analyzed (Participants) | 40 | 43 | 37
  Change at Week 8 | -10.01 (5.51) | -20.33 (5.20) | -7.28 (5.56)
Statistical Analysis 1: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.8633, ANCOVA; ANCOVA model with treatment, region, age group as terms, and Baseline score as a covariate for change from Baseline; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-12.48 to 10.48]
Statistical Analysis 2: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0452, ANCOVA; ANCOVA model with treatment, region, age group as terms, and Baseline score as a covariate for change from Baseline; Mean Difference (Final Values) = -11.54, 95% CI 2-sided [-22.83 to -0.25]
Statistical Analysis 3: Comparison: 0.3% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.6746, ANCOVA; ANCOVA model with treatment, region, age group as terms, and Baseline score as a covariate for change from Baseline; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-15.58 to 10.12]
Statistical Analysis 4: Comparison: 1% OPA-15406 vs Vehicle Ointment; Test type: Superiority or Other; p = 0.0432, ANCOVA; ANCOVA model with treatment, region, age group as terms, and Baseline score as a covariate for change from Baseline; Mean Difference (Final Values) = -13.05, 95% CI 2-sided [-25.69 to -0.4]

ADVERSE EVENTS:
Time Frame: From signing the informed consent until the end of the Treatment Period (Up to Week 8)
Description: Safety Sample included all participants who received at least one dose of IMP.
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406 | Vehicle Ointment
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/43 | 0/37
Serious Adverse Events (participants affected / at risk) | 2/41 | 2/43 | 0/37
Other Adverse Events (participants affected / at risk) | 22/41 | 13/43 | 16/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3% OPA-15406 (N=41) | 1% OPA-15406 (N=43) | Vehicle Ointment (N=37)
Giardiasis (Infections and infestations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3% OPA-15406 (N=41) | 1% OPA-15406 (N=43) | Vehicle Ointment (N=37)
Toothache (Gastrointestinal disorders) | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 3 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 11 | 7 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.